CLINICAL TRIAL: NCT04655976
Title: A Randomized, Open Label Phase 2/3 Study Comparing Cobolimab + Dostarlimab + Docetaxel To Dostarlimab + Docetaxel To Docetaxel Alone In Participants With Advanced Non-small Cell Lung Cancer Who Have Progressed On Prior Anti-PD-(L)1 Therapy And Chemotherapy (COSTAR Lung)
Brief Title: Efficacy Comparison of Cobolimab + Dostarlimab + Docetaxel to Dostarlimab + Docetaxel to Docetaxel Alone in Participants With Advanced Non-small Cell Lung Cancer Who Have Progressed on Prior Anti-PD-(L)1 Therapy and Chemotherapy
Acronym: COSTAR Lung
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213410; 2020-003433-37 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: GSK4069889A; GSK4057190A; Cobolimab; Dostarlimab; Docetaxel; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dostarlimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving cobolimab+ dostarlimab+ docetaxel (Experimental)
  Interventions: Biological: Cobolimab; Biological: Dostarlimab; Drug: Docetaxel
- Participants receiving dostarlimab+ docetaxel (Experimental)
  Interventions: Biological: Dostarlimab; Drug: Docetaxel
- Participants receiving docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Cobolimab — Cobolimab will be administered.
  Arms: Participants receiving cobolimab+ dostarlimab+ docetaxel
Biological: Dostarlimab — Dostarlimab will be administered.
  Arms: Participants receiving cobolimab+ dostarlimab+ docetaxel; Participants receiving dostarlimab+ docetaxel
Drug: Docetaxel — Docetaxel will be administered.

SUMMARY:
This is a multi-center, parallel group treatment, Phase 2/3 open label study evaluating cobolimab in combination with dostarlimab and docetaxel in participants with advanced non-small cell Lung Cancer (NSCLC) who have progressed on prior anti-PD-(L)1 therapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically proven advanced or metastatic NSCLC and only squamous or non-squamous cell carcinoma.
* Participant has received no more than 2 prior lines of therapy for advanced or metastatic disease, which must only include a platinum based (e.g., cisplatin, carboplatin) doublet chemotherapy regimen and an anti-PD-1 or an anti-PD-(L)1 antibody.
* Participant has measurable disease.
* Participant has documented radiographic disease progression on prior platinum based chemotherapy and on or after prior anti-PD-(L)1 therapy.
* Participant agrees to submit an archival formalin-fixed paraffin-embedded (FFPE) tumor tissue specimen that was collected on or after diagnosis of metastatic disease. If archival tissue is not available, the participant must undergo biopsy prior to study entry.
* Participant has an ECOG performance status score of 0 or 1.
* Participant has a life expectancy of at least 3 months.
* Participant has adequate Baseline organ function.
* Participant has recovered from any prior treatment related toxicities.
* Participant agrees to use contraception.

Exclusion Criteria:

* Participant has been previously treated with an anti-PD-[L]1 or anti-programmed death-ligand 2 (anti-PD-[L]2) agent that resulted in permanent discontinuation due to an AE.
* Participant has been previously treated with an anti-T cell immunoglobulin and mucin domain containing 3 (anti-TIM-3) or anti-cytotoxic T lymphocyte associated protein 4 (CTLA 4) agent or docetaxel.
* Participant has a documented sensitizing epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or c-ros oncogene 1 (ROS-1) mutation. Participants whose tumors have not been tested for these driver mutations and therefore who have unknown driver mutation status are not eligible. Participants with squamous histology do not need to be tested for these driver mutations.
* Participant had radiological or clinical disease progression (i.e., worsening performance status, clinical symptoms, and laboratory data) <=8 weeks after initiation of prior anti-programmed cell death protein 1 (anti-PD-1) or anti-PD-L1 antibody. The clinical disease progression should have been confirmed by a subsequent radiological scan.
* Participant has received radiation to the lung that is >30 gray (Gy) within 6 months prior to the first dose of study treatment.
* Participant has completed palliative radiotherapy within 7 days prior to the first dose of study treatment.
* Participant is ineligible if any of the following hepatic characteristics are present: a. Alanine aminotransferase (ALT) >2.5 times upper limit normal (ULN) b. ALT and/or aspartate aminotransferase (AST) >1.5 times ULN concomitant with alkaline phosphatase (ALP) >2.5 times ULN; c. Bilirubin >1 times ULN; d. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per the Investigator's assessment).
* Participant has known new or progressive brain metastases and/or leptomeningeal metastases. Participants who have received prior therapy for their brain metastases and have radiographically stable central nervous system disease may participate, provided they are neurologically stable for at least 4 weeks before study entry and are off corticosteroids within 3 days prior to the first dose of study treatment.
* Participant has tested positive for the following at Screening or within 3 months before the first dose of study treatment: a. Presence of hepatitis B surface antigen. b. Presence of hepatitis C antibody in the absence of a ribonucleic acid (RNA) test for hepatitis C virus. If a confirmatory RNA test is available, a positive test result will exclude a participant, while a negative test result (indicating absence of active infection) will allow the participant to enter into the study.
* Participant has known human immunodeficiency virus (HIV) (positive for HIV 1 or HIV 2 antibodies).
* Participant has active autoimmune disease that required systemic treatment in the past 2 years, is immunocompromised in the opinion of the Investigator, or is receiving systemic immunosuppressive treatment.
* Participant has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment of these conditions (including therapeutic thoracentesis or paracentesis) is eligible.
* Participant has current interstitial lung disease, current pneumonitis, or a history of pneumonitis that required the use of glucocorticoids to assist with management.
* Participant has pre-existing peripheral neuropathy that is Grade >=2 by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 criteria.
* Participant has received a live vaccine within 30 days of the first dose of study treatment. Seasonal flu vaccines that do not contain live virus and Coronavirus Disease 2019 (COVID-19) vaccines.
* Participant is unable to interrupt aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) for undergoing a biopsy procedure (in cases when a participant does not have an archival biopsy), other than an aspirin dose <=1.3 grams (g) per day, for a 5-day period (8-day) period for long-acting agents, such as piroxicam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in participants receiving cobolimab + dostarlimab + docetaxel relative to participants receiving docetaxel alone | Up to approximately 52 months
  OS is defined as survival from the date of randomization to the date of death by any cause.
OS in participants receiving dostarlimab + docetaxel relative to participants receiving docetaxel alone | Up to approximately 52 months
  OS is defined as survival from the date of randomization to the date of death by any cause.

SECONDARY OUTCOMES:
OS in participants receiving cobolimab + dostarlimab + docetaxel relative to participants receiving dostarlimab + docetaxel | Up to approximately 52 months
  OS is defined as survival from the date of randomization to the date of death by any cause.
Objective response rate (ORR) | Up to approximately 52 months
  Confirmed ORR is defined as the proportion of participants who have achieved confirmed complete response (CR) or confirmed partial response (PR), evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 based on Investigator assessment.
Progression free survival (PFS) | Up to approximately 52 months
  PFS is defined as the length of time until disease progression, from the time of randomization to the earliest date of assessment of disease progression based on RECIST version 1.1 by Investigator assessment or death by any cause.
Duration of response (DOR) | Up to approximately 52 months
  DOR is defined as the time from first documented response (CR/PR) until the time of first documentation of disease progression based on RECIST version 1.1 by Investigator assessment or death, whichever occurs first.
Time to deterioration (TTD) | Up to approximately 52 months
  TTD in lung cancer is defined as time from randomization to meaningful deterioration on a composite endpoint of dyspnea, chest pain, and cough, from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 13 item Lung Cancer Module (EORTC QLQ LC13).
Change from Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30 item Core Module (EORTC QLQ-C30) assessment | Baseline (Day 1) and up to approximately 52 months
  EORTC QLQ-C30 is a questionnaire used to measure health related quality of life (HRQoL) in participants with cancer.
Change from Baseline in the EORTC QLQ LC13 assessment | Baseline (Day 1) and up to approximately 52 months
  EORTC QLQ LC13 is a lung cancer specific questionnaire module designed to supplement the EORTC QLQ C30.
Number of participants with serious adverse events (SAEs) | From consent signature (Day -28) until the 90 day post last dose follow-up
Number of participants with treatment-emergent adverse events (TEAEs) and immune related adverse event (irAEs) | From consent signature (Day -28) until the 30 day post last dose follow-up
Number of participants with TEAEs leading to death | From consent signature (Day -28) until the 90 day post last dose follow-up
Number of participants with adverse events (AEs) leading to discontinuation | From consent signature (Day -28) until the 30 day post last dose follow-up
Number of participants with clinically significant changes in hematology, clinical chemistry, thyroid function and urinalysis lab parameters | From consent signature (Day -28) until the 90 day post last dose follow-up
  Blood and urine samples will be collected for the assessment of hematology, clinical chemistry, thyroid function and urinalysis lab parameters
Number of participants with clinically significant changes in vital signs and Electrocardiogram (ECG) Parameters | From consent signature (Day -28) until the 90 day post last dose follow-up
Number of participants with indicated Eastern Cooperative Oncology Group (ECOG) performance status | From consent signature (Day -28) until the 90 day post last dose follow-up
  Performance status will be assessed using the ECOG performance status scale. Scales range from grade 0 to 4, grade 0 denoting fully active and grade 4 completely disabled.
Number of participants with usage of concomitant medications | From consent signature (Day -28) until the 90 day post last dose follow-up
Number of participants with abnormal physical examinations | From consent signature (Day -28) until the 90 day post last dose follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (141):
- United States (16):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Edgewood, Kentucky
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, White Plains, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Tacoma, Washington
- Argentina (8):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Rioja
  - GSK Investigational Site, Pergamino
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Viedma
- Australia (6):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Ashford, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Ballarat, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Mount Waverley, Victoria
- Belgium (3):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Kortrijk
- Brazil (6):
  - GSK Investigational Site, Blumenau
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Canada (5):
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
- France (7):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Quimper
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Tours
- Germany (13):
  - GSK Investigational Site, Augsburg
  - GSK Investigational Site, Bad Berka
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Karlsruhe
  - GSK Investigational Site, München
  - GSK Investigational Site, Oldenburg
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Pylaia Thessaloniki
  - GSK Investigational Site, Rio Patras
  - GSK Investigational Site, Thessaloniki
- Italy (9):
  - GSK Investigational Site, Ancona
  - GSK Investigational Site, Avellino
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Orbassano to
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Siena
- Japan (4):
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Yamaguchi
- Mexico (4):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Puebla Puebla
- Netherlands (7):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zwolle
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Piła
  - GSK Investigational Site, Poznan
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Craiova Dolj
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Timișoara
- Russia (4):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow Region
  - GSK Investigational Site, Pushkin
  - GSK Investigational Site, Saint Petersburg
- South Korea (7):
  - GSK Investigational Site, Cheongju Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
- Spain (9):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gävle
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- GSK Investigational Site, Taipei, Taiwan
- Thailand (4):
  - GSK Investigational Site, Dusit
  - GSK Investigational Site, Kho Hong Hat Yai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Pathum Thani
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Izmir
- United Kingdom (4):
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com